CLINICAL TRIAL: NCT02915575
Title: Advancing Community Care and Access to Follow-up After Acute Kidney Injury Hospitalization
Brief Title: Improving Post Discharge Care After Acute Kidney Injury
Acronym: AFTER AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00067815
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (usual care) (Other): Participants will be discharged as per usual ward discharge protocols.
  Interventions: Other: Usual Care
- Risk guided follow-up (Other): Participant will be stratified for risk of CKD in three groups: Low (<1% risk of CKD), medium (1-10 % risk of CKD) and high (≥10 % risk of CKD). Specific follow-up will be guided by risk status
  Interventions: Other: Risk guided follow-up

INTERVENTIONS:
Other: Risk guided follow-up — Participant will be stratified for risk of CKD in three groups: Low (<1% risk of CKD), medium (1-10 % risk of CKD) and high (≥10 % risk of CKD). Specific follow-up will be guided by risk status
  Arms: Risk guided follow-up
Other: Usual Care — Participants will be discharged as per usual ward discharge protocols.
  Arms: Control Arm (usual care)

SUMMARY:
The purpose of this trial is to test the clinical benefit and feasibility of structured risk based post discharge care for hospital acquired Acute kidney injury survivors.This is a Pragmatic randomized controlled trial. It will be conducted at 2 hospitals in Alberta. 166 participants will be enrolled in this Randomized controlled trial..

DETAILED DESCRIPTION:
Research Objective:

To evaluate the impact of risk based decision support on processes of care for high-risk patients following discharge after hospitalization with Acute Kidney injury.

Experimental Strategy- rationale and considerations:

International guidelines for Chronic Kidney disease diagnosis and management provide a stage-based management approach to reduce the risk of adverse cardiovascular and renal outcomes based on estimated glomerular filtration rate (eGFR) and proteinuria. Identified key quality indicators for CKD care include the use of statins in CKD patients greater than age 50, or with diabetes or cardiovascular disease, use of ACEi (angiotensin-converting enzyme inhibitor) and ARB (angiotensin receptor blocker) in patients with proteinuria and referral to nephrology care with a sustained eGFR <30/ml/min/1.73m2. patients at low risk of CKD can be effectively managed by primary care given appropriate support. Study investigator will evaluate the identification of CKD by providing lab requisitions to all study participants. Those in the medium and high risk groups for CKD based on our risk index will be further guided to either a primary care web-based CKD care pathway which helps Primary care Physicians identify, treat and refer CKD patients using best practices, or nephrology care, respectively. Transitional care interventions have been shown to be effective preventing readmission in chronic conditions such as heart failure. Specialist care delivery often through multidisciplinary clinics has been found to improve prescription of proven efficacious medications and outcomes in a number of chronic disease settings including heart failure, Myocardial infarction,asthma and CKD. As there is no specific intervention for treating Acute kidney injury ensuring high adherence to CKD care in affected individuals is a feasible, sustainable strategy.

Participants The trial population will be comprised of consenting adult patients admitted to general medical or surgical teaching wards at 2 centers, the University of Alberta Hospital in Edmonton and the Foothills Hospital in Calgary.

Randomization

Participants will be randomized to either Control arm or Experimental arm

Control arm (Usual Care): Participants will be discharged as per usual ward discharge protocols. A requisition for follow-up labs (serum creatinine, serum electrolytes, urine albumin/creatinine ratio) to be drawn at 90 days will be given to each participant. Appointments/referrals will be left at the discretion of the care team.

Experimental arm (Risk Guided Follow-up): Participants will be stratified for risk of CKD into three groups: low (<1% risk of CKD), medium (1-10 % risk of CKD) and high (≥10 % risk of CKD) using a risk index developed by the team. Specific follow-up will be guided by risk status.

Analysis Plan:

The primary analysis will follow an intention-to-treat approach. In sensitivity analyses, outcomes based on the predicted risk of CKD will be stratified. Descriptive statistics and bivariate tests of associations will be used as appropriate to evaluate group differences at various time points of follow-up. Associations between key variables and study outcomes will be analyzed using appropriate univariate, multivariate and mixed model multilevel analyses. No interim analyses are planned due to the short duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yrs
* At least a doubling of serum creatinine during hospitalization (including need for dialysis)
* Have a primary care physician (PCP)
* No nephrologist follow up arranged after hospital discharge

Exclusion Criteria:

* Baseline GFR<30ml/min/1.73m2(CKD-EPI) or requiring chronic dialysis on admission
* Renal transplant recipients
* Poor prognosis not expected to survive > 6 months
* Residence at a nursing home facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients develop Chronic kidney disease after Acute kidney injury | 90 days
  The primary (process based) outcome of this trial is the proportion of patients with CKD meeting all three quality of care indicators (statin use, ACEi/ARB use in those with proteinuria (ACR>30mg/mmol) or diabetes, nephrologist visit if sustained eGFR<30ml/min/1.73m2) within 90 days of hospital

SECONDARY OUTCOMES:
Proportion of patients completed the lab and seen by PCP | 90 days
  Participant discharged from the hospital will be given lab requisition, to be drawn within 90 days
check eGFR | one year
  Participant will have their eGFR check at one year
Hospitalization | one year
  Proportion of patients hospitalized for AKI or renal specific condition
Feasibility | one year
  Proportion of eligible patients recruited in the study

CONTACTS AND LOCATIONS:
Overall Officials: Neesh Pannu, MD, Principal Investigator — University of Alberta; Matthew James, MD, Principal Investigator — Foothills Medical Centre
Locations (2):
- Canada (2):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No